CLINICAL TRIAL: NCT01219725
Title: Can a Moderate Intensity Exercise Training Programme Improve Cardiac Function and Known Cardiovascular Risk Factors in Middle-aged Women?
Brief Title: Cardiovascular Prophylaxis for Postmenopausal Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Dr Karen Michelle Birch, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RG2508/06/08
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2009-05

CONDITIONS: Cardiovascular Disease
Keywords: Body composition; Endothelial function; Lipoprotein profile; Inflammatory markers; Aerobic capacity; Thrombotic markers; Arterial stiffness; Cardiac function; Traditional and emerging cardiovascular disease risk factors
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Exercise training — 6 months of moderate intensity exercise training 3 times per week

SUMMARY:
The purpose of this study was to examine the effect of 6 months moderate intensity exercise training completed three times per week upon traditional and emerging cardiovascular disease risk factors in postmenopausal women both with and without type 2 diabetes. These risk factors include blood markers associated with increased risk such as cholesterol, insulin, glucose and markers of inflammation plus measures of body fat, heart and lung fitness, vascular stiffness and vascular function. The study hypothesised that moderate intensity exercise training would intervene in the exaggerated risk seen in women following the menopause, especially in those with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and stable type II diabetic postmenopausal women (cessation of menstrual periods for 12 months and confirmed with LH/FSH samples) aged 45 - 65 years old for the cross sectional analysis and exercise training study.

Exclusion Criteria:

* Identified abnormalities during baseline testing.
* Vigorously active women.
* Women who are pregnant.
* Women with serious systemic or psychological disorders (e.g. COPD, asthma, clinical depression).
* Women with known coronary artery disease.
* Women with significant cardiovascular pathologies and associated medication.
* Women with type 1 or insulin treated diabetes.
* Women with diabetes with complications.
* Women with unstable diabetes or hypertension.
* Women with any cancer.
* Women with musculoskeletal impairments or contraindications to exercise.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake | 6 months

SECONDARY OUTCOMES:
lipoprotein profile | 6 months
Flow mediated dilation | 6 months
Cardiac power output | 6 months
Arterial stiffness | 6 months
Inflammatory markers | 6 months
Body composition | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Birch, BSC, PhD, Principal Investigator — University of Leeds
Locations (1):
- Centre for Sports and Exercise Sciences, University of Leeds, Leeds, West Yorkshire, United Kingdom